CLINICAL TRIAL: NCT01179048
Title: A Long-term, Multi-centre, International, Randomised Double-blind, Placebo-controlled Trial to Determine Liraglutide Effects on Cardiovascular Events
Brief Title: Liraglutide Effect and Action in Diabetes: Evaluation of Cardiovascular Outcome Results
Acronym: LEADER®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EX2211-3748; 2009-012201-19 (EudraCT Number); U1111-1113-7090 (Other: WHO); CTR20130003 (Other: CFDA)
Record Dates: First submitted 2010-08-06; First posted 2010-08-10 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Maximum dose of 1.8 mg liraglutide, injected subcutaneously (under the skin) once daily. Administered in addition to the subject's standard treatment
  Arms: Liraglutide
Drug: placebo — Maximum dose of 1.8 mg placebo, injected subcutaneously (under the skin) once daily. Administered in addition to the subject's standard treatment
  Arms: Placebo

SUMMARY:
This trial is conducted in Africa, Asia, Europe, and North and South America. The aim of this trial is to determine the long term effect of liraglutide on cardiovascular events in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria: - Type 2 diabetes - Age min. 50 years at screening and concomitant cardiovascular, cerebrovascular or peripheral vascular disease or chronic renal failure or chronic heart failure OR age min. 60 years at screening and other specified risk factors of cardiovascular disease - HbA1c: 7.0% or above - Anti-diabetic drug naive or treated with one or more oral anti-diabetic drugs (OADs) or treated with human NPH insulin or long-acting insulin analogue or premixed insulin, alone or in combination with OAD(s) Exclusion Criteria: - Type 1 diabetes - Use of a glucagon-like peptide-1 (GLP-1) receptor agonist (exenatide, liraglutide or other) or pramlintide or any dipeptidyl peptidase 4 (DPP-4) inhibitor within the 3 months prior to screening (trial start) - Use of insulin other than human NPH insulin or long-acting insulin analogue or premixed insulin within 3 months prior to screening. Short-term use of other insulin during this period in connection with intercurrent illness is allowed, at Investigator's discretion

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9341 (Actual)
Dates: Start 2010-08-31 (Actual); Primary Completion 2015-12-17 (Actual); Study Completion 2015-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (352):
- United States (109):
  - Novo Nordisk Investigational Site, Alabaster, Alabama
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Huntsville, Alabama
  - Novo Nordisk Investigational Site, Mobile, Alabama
  - Novo Nordisk Investigational Site, Tempe, Arizona
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Cerritos, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Los Banos, California
  - Novo Nordisk Investigational Site, Mission Hills, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Watsonville, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Newark, Delaware
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, DeLand, Florida
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Crystal Lake, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Michigan City, Indiana
  - Novo Nordisk Investigational Site, West Des Moines, Iowa
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Monroe, Louisiana
  - Novo Nordisk Investigational Site, Natchitoches, Louisiana
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Bloomfield Hills, Michigan
  - Novo Nordisk Investigational Site, Dearborn, Michigan
  - Novo Nordisk Investigational Site, Interlochen, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Springfield, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Great Falls, Montana
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Lebanon, New Hampshire
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Mine Hill, New Jersey
  - Novo Nordisk Investigational Site, Neptune City, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Smithtown, New York
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, Westfield, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Burlington, North Carolina
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Monroe, North Carolina
  - Novo Nordisk Investigational Site, Mooresville, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Cadiz, Ohio
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Marion, Ohio
  - Novo Nordisk Investigational Site, Middleburg Heights, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Hatfield, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Uniontown, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Columbia, South Carolina
  - Novo Nordisk Investigational Site, Greenville, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Murrells Inlet, South Carolina
  - Novo Nordisk Investigational Site, Myrtle Beach, South Carolina
  - Novo Nordisk Investigational Site, Bartlett, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Longview, Texas
  - Novo Nordisk Investigational Site, Lubbock, Texas
  - Novo Nordisk Investigational Site, Odessa, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Schertz, Texas
  - Novo Nordisk Investigational Site, Tomball, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, South Burlington, Vermont
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Madison, Wisconsin
- Australia (10):
  - Novo Nordisk Investigational Site, Blacktown, New South Wales
  - Novo Nordisk Investigational Site, Douglas, Queensland
  - Novo Nordisk Investigational Site, Herston, Queensland
  - Novo Nordisk Investigational Site, Meadowbrook, Queensland
  - Novo Nordisk Investigational Site, Keswick, South Australia
  - Novo Nordisk Investigational Site, Oaklands Park, South Australia
  - Novo Nordisk Investigational Site, Hobart, Tasmania
  - Novo Nordisk Investigational Site, Box Hill, Victoria
  - Novo Nordisk Investigational Site, Fitzroy, Victoria
  - Novo Nordisk Investigational Site, Fremantle, Western Australia
- Austria (2):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Vienna
- Belgium (4):
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Ghent
  - Novo Nordisk Investigational Site, Leuven
  - Novo Nordisk Investigational Site, Liège
- Brazil (22):
  - Novo Nordisk Investigational Site, Fortaleza, Ceará
  - Novo Nordisk Investigational Site, Aparecida de Goiânia, Goiás
  - Novo Nordisk Investigational Site, Curitiba, Paraná
  - Novo Nordisk Investigational Site, Belém, Pará
  - Novo Nordisk Investigational Site, Caxias do Sul, Rio Grande do Sul
  - Novo Nordisk Investigational Site, Porto Alegre, Rio Grande do Sul
  - Novo Nordisk Investigational Site, Campinas, São Paulo
  - Novo Nordisk Investigational Site, Mogi das Cruzes, São Paulo
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Aracajú
  - Novo Nordisk Investigational Site, Belo Horizonte
  - Novo Nordisk Investigational Site, Campinas
  - Novo Nordisk Investigational Site, Curitiba
  - Novo Nordisk Investigational Site, Fortaleza
  - Novo Nordisk Investigational Site, Goiânia
  - Novo Nordisk Investigational Site, Joinville
  - Novo Nordisk Investigational Site, Marília
  - Novo Nordisk Investigational Site, Porto Alegre
  - Novo Nordisk Investigational Site, Recife
  - Novo Nordisk Investigational Site, Rio de Janeiro
  - Novo Nordisk Investigational Site, Santos
  - Novo Nordisk Investigational Site, São Paulo
- Canada (15):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, St. John's, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Cambridge, Ontario
  - Novo Nordisk Investigational Site, Cornwall, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Mississauga, Ontario
  - Novo Nordisk Investigational Site, Scarborough Village, Ontario
  - Novo Nordisk Investigational Site, Smiths Falls, Ontario
  - Novo Nordisk Investigational Site, Thunder Bay, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Québec
- China (6):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Xiamen, Fujian
  - Novo Nordisk Investigational Site, Guangzhou, Guangdong
  - Novo Nordisk Investigational Site, Zhenjiang, Jiangsu
  - Novo Nordisk Investigational Site, Qingdao, Shandong
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
- Czechia (2):
  - Novo Nordisk Investigational Site, Pilsen
  - Novo Nordisk Investigational Site, Prague
- Denmark (6):
  - Novo Nordisk Investigational Site, Aalborg
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Esbjerg
  - Novo Nordisk Investigational Site, Gentofte Municipality
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, Odense
- Finland (5):
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Lahti
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Vantaa
- France (4):
  - Novo Nordisk Investigational Site, Corbeil-Essonnes
  - Novo Nordisk Investigational Site, Jarny
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Paris
- Germany (22):
  - Novo Nordisk Investigational Site, Angermünde/OT Wolletz
  - Novo Nordisk Investigational Site, Aschaffenburg
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Dillingen
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Elsterwerda
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Gifhorn
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Karlsbad
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Mannheim
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Oldenburg
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Schkeuditz
  - Novo Nordisk Investigational Site, Schweinfurt
  - Novo Nordisk Investigational Site, Ulm
  - Novo Nordisk Investigational Site, Villingen-Schwenningen
  - Novo Nordisk Investigational Site, Wangen
- Greece (3):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Crete
  - Novo Nordisk Investigational Site, Thessaloniki
- India (15):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Hyderbad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Guwahati, Assam
  - Novo Nordisk Investigational Site, Karnāl, Haryana
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Manipal, Karnataka
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Chandigarh, Punjab
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Madurai, Tamil Nadu
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Thriruvananthapuram
- Novo Nordisk Investigational Site, Dublin, Ireland
- Israel (4):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Italy (10):
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Chieti
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Latina
  - Novo Nordisk Investigational Site, Lucca
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Roma
- Mexico (6):
  - Novo Nordisk Investigational Site, Tijuana, Baja California Norte
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Aguascalientes
  - Novo Nordisk Investigational Site, Durango
  - Novo Nordisk Investigational Site, Monterrey
  - Novo Nordisk Investigational Site, San Luis Potosí City
- Netherlands (9):
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Etten-Leur
  - Novo Nordisk Investigational Site, Goes
  - Novo Nordisk Investigational Site, Groningen
  - Novo Nordisk Investigational Site, Hoogeveen
  - Novo Nordisk Investigational Site, Maastricht
  - Novo Nordisk Investigational Site, Nijmegen
  - Novo Nordisk Investigational Site, Utrecht
- Norway (4):
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Trondheim
  - Novo Nordisk Investigational Site, Tønsberg
- Poland (10):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Bydgoszcz
  - Novo Nordisk Investigational Site, Katowice
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Puławy
  - Novo Nordisk Investigational Site, Ruda Śląska
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Puerto Rico (2):
  - Novo Nordisk Investigational Site, Bayamón
  - Novo Nordisk Investigational Site, Caguas
- Romania (10):
  - Novo Nordisk Investigational Site, Craiova, Dolj
  - Novo Nordisk Investigational Site, Târgu Mureş, Mureș County
  - Novo Nordisk Investigational Site, Timișoara, Timiș County
  - Novo Nordisk Investigational Site, Bacau
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Constanța
  - Novo Nordisk Investigational Site, Deva
  - Novo Nordisk Investigational Site, Iași
  - Novo Nordisk Investigational Site, Satu Mare
  - Novo Nordisk Investigational Site, Sibiu
- Russia (10):
  - Novo Nordisk Investigational Site, Arkhangelsk
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Nizhny Novgorod
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Smolensk
  - Novo Nordisk Investigational Site, Tyumen
  - Novo Nordisk Investigational Site, Yaroslavl
- Novo Nordisk Investigational Site, Belgrade, Serbia
- South Africa (11):
  - Novo Nordisk Investigational Site, Bloemfontein, Free State
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Lenasia, Gauteng
  - Novo Nordisk Investigational Site, Midrand, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Tongaat, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
  - Novo Nordisk Investigational Site, Somerset West, Western Cape
  - Novo Nordisk Investigational Site, Alberton
  - Novo Nordisk Investigational Site, Cape Town
- South Korea (3):
  - Novo Nordisk Investigational Site, Goyang
  - Novo Nordisk Investigational Site, Seongnam-si
  - Novo Nordisk Investigational Site, Seoul
- Spain (10):
  - Novo Nordisk Investigational Site, A Coruña
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Mora de Ebre
  - Novo Nordisk Investigational Site, Mostoles - Madrid -
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Pozuelo de Alarcón
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valladolid
- Sweden (4):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Örebro
  - Novo Nordisk Investigational Site, Stockholm
- Taiwan (4):
  - Novo Nordisk Investigational Site, Changhua
  - Novo Nordisk Investigational Site, Kaoshiung
  - Novo Nordisk Investigational Site, Tainan
  - Novo Nordisk Investigational Site, Taoyuan District
- Turkey (Türkiye) (7):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Bursa
  - Novo Nordisk Investigational Site, Gaziantep
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir
  - Novo Nordisk Investigational Site, Kayseri
- Novo Nordisk Investigational Site, Dubai, United Arab Emirates
- United Kingdom (20):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Devon
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Livington
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Norwich
  - Novo Nordisk Investigational Site, Nuneaton
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, St Helens
  - Novo Nordisk Investigational Site, Swansea
  - Novo Nordisk Investigational Site, Torquay
  - Novo Nordisk Investigational Site, West Midlands

REFERENCES:
- [Background] Verma S, Bain SC, Monk Fries T, Mazer CD, Nauck MA, Pratley RE, Rasmussen S, Saevereid HA, Zinman B, Buse JB. Duration of diabetes and cardiorenal efficacy of liraglutide and semaglutide: A post hoc analysis of the LEADER and SUSTAIN 6 clinical trials. Diabetes Obes Metab. 2019 Jul;21(7):1745-1751. doi: 10.1111/dom.13698. Epub 2019 Apr 2. PMID 30851070
- [Background] Hinton W, Feher M, Munro N, Walker M, de Lusignan S. Real-world prevalence of the inclusion criteria for the LEADER trial: Data from a national general practice network. Diabetes Obes Metab. 2019 Jul;21(7):1661-1667. doi: 10.1111/dom.13710. Epub 2019 Apr 11. PMID 30900349
- [Result] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Result] Petrie JR, Marso SP, Bain SC, Franek E, Jacob S, Masmiquel L, Leiter LA, Haluzik M, Satman I, Omar M, Shestakova M, Van Gaal L, Mann JF, Baeres FM, Zinman B, Poulter NR; LEADER investigators. LEADER-4: blood pressure control in patients with type 2 diabetes and high cardiovascular risk: baseline data from the LEADER randomized trial. J Hypertens. 2016 Jun;34(6):1140-50. doi: 10.1097/HJH.0000000000000890. PMID 26855018
- [Result] Masmiquel L, Leiter LA, Vidal J, Bain S, Petrie J, Franek E, Raz I, Comlekci A, Jacob S, van Gaal L, Baeres FM, Marso SP, Eriksson M; LEADER investigators. LEADER 5: prevalence and cardiometabolic impact of obesity in cardiovascular high-risk patients with type 2 diabetes mellitus: baseline global data from the LEADER trial. Cardiovasc Diabetol. 2016 Feb 10;15:29. doi: 10.1186/s12933-016-0341-5. PMID 26864124
- [Result] Satman I, R Rea R, Eriksson M, Mosenzon O, Pratley R, M Baeres F, D Orsted D, F Mann J; LEADER Trial Investigators. LEADER-6: Baseline renal function and associated factors in a high cardiovascular risk type 2 diabetes population. J Diabetes Complications. 2016 Nov-Dec;30(8):1631-1639. doi: 10.1016/j.jdiacomp.2016.06.001. Epub 2016 Jun 3. PMID 27320184
- [Result] Rutten GE, Tack CJ, Pieber TR, Comlekci A, Orsted DD, Baeres FM, Marso SP, Buse JB; LEADER Investigators. LEADER 7: cardiovascular risk profiles of US and European participants in the LEADER diabetes trial differ. Diabetol Metab Syndr. 2016 Jun 2;8:37. doi: 10.1186/s13098-016-0153-5. eCollection 2016. PMID 27274772
- [Result] Marso SP, Poulter NR, Nissen SE, Nauck MA, Zinman B, Daniels GH, Pocock S, Steinberg WM, Bergenstal RM, Mann JF, Ravn LS, Frandsen KB, Moses AC, Buse JB. Design of the liraglutide effect and action in diabetes: evaluation of cardiovascular outcome results (LEADER) trial. Am Heart J. 2013 Nov;166(5):823-30.e5. doi: 10.1016/j.ahj.2013.07.012. Epub 2013 Oct 2. PMID 24176437
- [Result] Steinberg WM, Nauck MA, Zinman B, Daniels GH, Bergenstal RM, Mann JF, Steen Ravn L, Moses AC, Stockner M, Baeres FM, Marso SP, Buse JB; LEADER Trial investigators. LEADER 3--lipase and amylase activity in subjects with type 2 diabetes: baseline data from over 9000 subjects in the LEADER Trial. Pancreas. 2014 Nov;43(8):1223-31. doi: 10.1097/MPA.0000000000000229. PMID 25275271
- [Result] Daniels GH, Hegedus L, Marso SP, Nauck MA, Zinman B, Bergenstal RM, Mann JF, Derving Karsbol J, Moses AC, Buse JB, Tuttle RM; LEADER Trial Investigators. LEADER 2: baseline calcitonin in 9340 people with type 2 diabetes enrolled in the Liraglutide Effect and Action in Diabetes: Evaluation of cardiovascular outcome Results (LEADER) trial: preliminary observations. Diabetes Obes Metab. 2015 May;17(5):477-86. doi: 10.1111/dom.12444. Epub 2015 Feb 23. PMID 25656058
- [Result] Steinberg WM, Buse JB, Ghorbani MLM, Orsted DD, Nauck MA; LEADER Steering Committee; LEADER Trial Investigators. Amylase, Lipase, and Acute Pancreatitis in People With Type 2 Diabetes Treated With Liraglutide: Results From the LEADER Randomized Trial. Diabetes Care. 2017 Jul;40(7):966-972. doi: 10.2337/dc16-2747. Epub 2017 May 5. PMID 28476871
- [Result] Mann JFE, Orsted DD, Brown-Frandsen K, Marso SP, Poulter NR, Rasmussen S, Tornoe K, Zinman B, Buse JB; LEADER Steering Committee and Investigators. Liraglutide and Renal Outcomes in Type 2 Diabetes. N Engl J Med. 2017 Aug 31;377(9):839-848. doi: 10.1056/NEJMoa1616011. PMID 28854085
- [Result] Hegedus L, Sherman SI, Tuttle RM, von Scholten BJ, Rasmussen S, Karsbol JD, Daniels GH; LEADER Publication Committee on behalf of the LEADER Trial Investigators. No Evidence of Increase in Calcitonin Concentrations or Development of C-Cell Malignancy in Response to Liraglutide for Up to 5 Years in the LEADER Trial. Diabetes Care. 2018 Mar;41(3):620-622. doi: 10.2337/dc17-1956. Epub 2017 Dec 26. PMID 29279300
- [Result] Marso SP, Nauck MA, Monk Fries T, Rasmussen S, Treppendahl MB, Buse JB; LEADER Publication Committee on behalf of the LEADER Trial Investigators. Myocardial Infarction Subtypes in Patients With Type 2 Diabetes Mellitus and the Effect of Liraglutide Therapy (from the LEADER Trial). Am J Cardiol. 2018 Jun 15;121(12):1467-1470. doi: 10.1016/j.amjcard.2018.02.030. Epub 2018 Mar 15. PMID 29627109
- [Result] Verma S, Bhatt DL, Bain SC, Buse JB, Mann JFE, Marso SP, Nauck MA, Poulter NR, Pratley RE, Zinman B, Michelsen MM, Monk Fries T, Rasmussen S, Leiter LA; LEADER Publication Committee on behalf of the LEADER Trial Investigators. Effect of Liraglutide on Cardiovascular Events in Patients With Type 2 Diabetes Mellitus and Polyvascular Disease: Results of the LEADER Trial. Circulation. 2018 May 15;137(20):2179-2183. doi: 10.1161/CIRCULATIONAHA.118.033898. No abstract available. PMID 29760228
- [Result] Nauck MA, Jensen TJ, Rosenkilde C, Calanna S, Buse JB; LEADER Publication Committee on behalf of the LEADER Trial Investigators. Neoplasms Reported With Liraglutide or Placebo in People With Type 2 Diabetes: Results From the LEADER Randomized Trial. Diabetes Care. 2018 Aug;41(8):1663-1671. doi: 10.2337/dc17-1825. Epub 2018 Jun 13. PMID 29898902
- [Result] Zinman B, Marso SP, Christiansen E, Calanna S, Rasmussen S, Buse JB; LEADER Publication Committee on behalf of the LEADER Trial Investigators. Hypoglycemia, Cardiovascular Outcomes, and Death: The LEADER Experience. Diabetes Care. 2018 Aug;41(8):1783-1791. doi: 10.2337/dc17-2677. Epub 2018 Jun 14. PMID 29903847
- [Result] Nauck MA, Tornoe K, Rasmussen S, Treppendahl MB, Marso SP; LEADER Publication Committee on behalf of the LEADER Trial Investigators. Cardiovascular outcomes in patients who experienced a myocardial infarction while treated with liraglutide versus placebo in the LEADER trial. Diab Vasc Dis Res. 2018 Sep;15(5):465-468. doi: 10.1177/1479164118783935. Epub 2018 Jun 27. PMID 29947247
- [Result] Dhatariya K, Bain SC, Buse JB, Simpson R, Tarnow L, Kaltoft MS, Stellfeld M, Tornoe K, Pratley RE; LEADER Publication Committee on behalf of the LEADER Trial Investigators. The Impact of Liraglutide on Diabetes-Related Foot Ulceration and Associated Complications in Patients With Type 2 Diabetes at High Risk for Cardiovascular Events: Results From the LEADER Trial. Diabetes Care. 2018 Oct;41(10):2229-2235. doi: 10.2337/dc18-1094. Epub 2018 Aug 2. PMID 30072400
- [Result] Verma S, Leiter LA, Mazer CD, Bain SC, Buse J, Marso S, Nauck M, Zinman B, Bosch-Traberg H, Rasmussen S, Michelsen MM, Bhatt DL. Liraglutide Reduces Cardiovascular Events and Mortality in Type 2 Diabetes Mellitus Independently of Baseline Low-Density Lipoprotein Cholesterol Levels and Statin Use. Circulation. 2018 Oct 9;138(15):1605-1607. doi: 10.1161/CIRCULATIONAHA.118.036862. No abstract available. PMID 30354517
- [Result] Mann JFE, Fonseca V, Mosenzon O, Raz I, Goldman B, Idorn T, von Scholten BJ, Poulter NR. Effects of Liraglutide Versus Placebo on Cardiovascular Events in Patients With Type 2 Diabetes Mellitus and Chronic Kidney Disease. Circulation. 2018 Dec 18;138(25):2908-2918. doi: 10.1161/CIRCULATIONAHA.118.036418. PMID 30566006
- [Result] Verma S, Poulter NR, Bhatt DL, Bain SC, Buse JB, Leiter LA, Nauck MA, Pratley RE, Zinman B, Orsted DD, Monk Fries T, Rasmussen S, Marso SP. Effects of Liraglutide on Cardiovascular Outcomes in Patients With Type 2 Diabetes Mellitus With or Without History of Myocardial Infarction or Stroke. Circulation. 2018 Dec 18;138(25):2884-2894. doi: 10.1161/CIRCULATIONAHA.118.034516. PMID 30566004
- [Result] Nauck MA, Buse JB, Mann JFE, Pocock S, Bosch-Traberg H, Frimer-Larsen H, Ye Q, Gray A; LEADER Publication Committee for the LEADER Trial Investigators. Health-related quality of life in people with type 2 diabetes participating in the LEADER trial. Diabetes Obes Metab. 2019 Mar;21(3):525-532. doi: 10.1111/dom.13547. Epub 2018 Oct 25. PMID 30260088
- [Result] Zinman B, Nauck MA, Bosch-Traberg H, Frimer-Larsen H, Orsted DD, Buse JB; LEADER Publication Committee on behalf of the LEADER Trial Investigators. Liraglutide and Glycaemic Outcomes in the LEADER Trial. Diabetes Ther. 2018 Dec;9(6):2383-2392. doi: 10.1007/s13300-018-0524-z. Epub 2018 Nov 3. PMID 30392095
- [Result] Gilbert MP, Bain SC, Franek E, Jodar-Gimeno E, Nauck MA, Pratley R, Rea RR, Kerr Saraiva JF, Rasmussen S, Tornoe K, von Scholten BJ, Buse JB; LEADER Publication Committee on behalf of the LEADER Trial Investigators. Effect of Liraglutide on Cardiovascular Outcomes in Elderly Patients: A Post Hoc Analysis of a Randomized Controlled Trial. Ann Intern Med. 2019 Mar 19;170(6):423-426. doi: 10.7326/M18-1569. Epub 2018 Dec 4. No abstract available. PMID 30508430
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Verma S, Al-Omran M, Leiter LA, Mazer CD, Rasmussen S, Saevereid HA, Sejersten Ripa M, Bonaca MP. Cardiovascular efficacy of liraglutide and semaglutide in individuals with diabetes and peripheral artery disease. Diabetes Obes Metab. 2022 Jul;24(7):1288-1299. doi: 10.1111/dom.14700. Epub 2022 Apr 11. PMID 35332654
- [Derived] Heller SR, Geybels MS, Iqbal A, Liu L, Wagner L, Chow E. A higher non-severe hypoglycaemia rate is associated with an increased risk of subsequent severe hypoglycaemia and major adverse cardiovascular events in individuals with type 2 diabetes in the LEADER study. Diabetologia. 2022 Jan;65(1):55-64. doi: 10.1007/s00125-021-05556-7. Epub 2021 Oct 26. PMID 34704120
- [Derived] Persson F, Bain SC, Mosenzon O, Heerspink HJL, Mann JFE, Pratley R, Raz I, Idorn T, Rasmussen S, von Scholten BJ, Rossing P; LEADER Trial Investigators. Changes in Albuminuria Predict Cardiovascular and Renal Outcomes in Type 2 Diabetes: A Post Hoc Analysis of the LEADER Trial. Diabetes Care. 2021 Apr;44(4):1020-1026. doi: 10.2337/dc20-1622. Epub 2021 Jan 27. PMID 33504496
- [Derived] Verma S, McGuire DK, Bain SC, Bhatt DL, Leiter LA, Mazer CD, Monk Fries T, Pratley RE, Rasmussen S, Vrazic H, Zinman B, Buse JB. Effects of glucagon-like peptide-1 receptor agonists liraglutide and semaglutide on cardiovascular and renal outcomes across body mass index categories in type 2 diabetes: Results of the LEADER and SUSTAIN 6 trials. Diabetes Obes Metab. 2020 Dec;22(12):2487-2492. doi: 10.1111/dom.14160. Epub 2020 Sep 4. PMID 32744418
- [Derived] Crowley MJ, McGuire DK, Alexopoulos AS, Jensen TJ, Rasmussen S, Saevereid HA, Verma S, Buse JB. Effects of Liraglutide on Cardiovascular Outcomes in Type 2 Diabetes Patients With and Without Baseline Metformin Use: Post Hoc Analyses of the LEADER Trial. Diabetes Care. 2020 Sep;43(9):e108-e110. doi: 10.2337/dc20-0437. Epub 2020 Jul 9. No abstract available. PMID 32647053
- [Derived] Verma S, Bain SC, Honore JB, F E Mann J, A Nauck M, E Pratley R, Rasmussen S, Sejersten Ripa M, Zinman B, Buse JB. Impact of microvascular disease on cardiovascular outcomes in type 2 diabetes: Results from the LEADER and SUSTAIN 6 clinical trials. Diabetes Obes Metab. 2020 Nov;22(11):2193-2198. doi: 10.1111/dom.14140. Epub 2020 Aug 12. PMID 32643857
- [Derived] Leiter LA, Bain SC, Bhatt DL, Buse JB, Mazer CD, Pratley RE, Rasmussen S, Ripa MS, Vrazic H, Verma S. The effect of glucagon-like peptide-1 receptor agonists liraglutide and semaglutide on cardiovascular and renal outcomes across baseline blood pressure categories: Analysis of the LEADER and SUSTAIN 6 trials. Diabetes Obes Metab. 2020 Sep;22(9):1690-1695. doi: 10.1111/dom.14079. Epub 2020 Jun 3. PMID 32372454
- [Derived] Buse JB, Bain SC, Mann JFE, Nauck MA, Nissen SE, Pocock S, Poulter NR, Pratley RE, Linder M, Monk Fries T, Orsted DD, Zinman B; LEADER Trial Investigators. Cardiovascular Risk Reduction With Liraglutide: An Exploratory Mediation Analysis of the LEADER Trial. Diabetes Care. 2020 Jul;43(7):1546-1552. doi: 10.2337/dc19-2251. Epub 2020 May 4. PMID 32366578
- [Derived] Marso SP, Baeres FMM, Bain SC, Goldman B, Husain M, Nauck MA, Poulter NR, Pratley RE, Thomsen AB, Buse JB; LEADER Trial Investigators. Effects of Liraglutide on Cardiovascular Outcomes in Patients With Diabetes With or Without Heart Failure. J Am Coll Cardiol. 2020 Mar 17;75(10):1128-1141. doi: 10.1016/j.jacc.2019.12.063. PMID 32164886
- [Derived] Mann JFE, Fonseca VA, Poulter NR, Raz I, Idorn T, Rasmussen S, von Scholten BJ, Mosenzon O; LEADER Trial Investigators. Safety of Liraglutide in Type 2 Diabetes and Chronic Kidney Disease. Clin J Am Soc Nephrol. 2020 Apr 7;15(4):465-473. doi: 10.2215/CJN.11881019. Epub 2020 Mar 4. PMID 32132141
- [Derived] Nauck MA, Kreiner E, Rasmussen S, Saevereid HA, Buse JB; LEADER Trial Investigators. Response to Comment on Nauck et al. Effects of Liraglutide Compared With Placebo on Events of Acute Gallbladder or Biliary Disease in Patients With Type 2 Diabetes at High Risk for Cardiovascular Events in the LEADER Randomized Trial. Diabetes Care 2019;42:1912-1920. Diabetes Care. 2020 Feb;43(2):e30-e31. doi: 10.2337/dci19-0067. No abstract available. PMID 31959650
- [Derived] Verma S, Bain SC, Buse JB, Idorn T, Rasmussen S, Orsted DD, Nauck MA. Occurence of First and Recurrent Major Adverse Cardiovascular Events With Liraglutide Treatment Among Patients With Type 2 Diabetes and High Risk of Cardiovascular Events: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2019 Dec 1;4(12):1214-1220. doi: 10.1001/jamacardio.2019.3080. PMID 31721979
- [Derived] Nauck MA, Muus Ghorbani ML, Kreiner E, Saevereid HA, Buse JB; LEADER Publication Committee on behalf of the LEADER Trial Investigators. Effects of Liraglutide Compared With Placebo on Events of Acute Gallbladder or Biliary Disease in Patients With Type 2 Diabetes at High Risk for Cardiovascular Events in the LEADER Randomized Trial. Diabetes Care. 2019 Oct;42(10):1912-1920. doi: 10.2337/dc19-0415. Epub 2019 Aug 9. PMID 31399438
- [Derived] Tack CJ, Jacob S, Desouza C, Bain SC, Buse JB, Nauck MA, Petrie JR, Poulter NR, Pratley RE, Stegmann HVBK, Bosch-Traberg H, Startseva E, Zinman B; LEADER Publication Committee on behalf of the LEADER Trial Investigators. Long-term efficacy and safety of combined insulin and glucagon-like peptide-1 therapy: Evidence from the LEADER trial. Diabetes Obes Metab. 2019 Nov;21(11):2450-2458. doi: 10.1111/dom.13826. Epub 2019 Jul 7. PMID 31282028
- [Derived] Wittbrodt ET, Eudicone JM, Bell KF, Enhoffer DM, Latham K, Green JB. Generalizability of glucagon-like peptide-1 receptor agonist cardiovascular outcome trials enrollment criteria to the US type 2 diabetes population. Am J Manag Care. 2018 Apr;24(8 Suppl):S146-S155. PMID 29693361
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 410 sites in 32 countries across the 4 regions recruited subjects. Number of sites that recruited subjects is given in parenthesis. Europe (143), North America (135) (US, Canada) , Asia (33) (China, Taiwan, Korea, India) and Rest of the world (99) (Brazil, Mexico, Australia, South Africa, Turkey, Russian Federation, United Arab Emirates).
Pre-assignment Details: All subjects received placebo (0.6 mg/day) during the open labeled run-in period of 2-3 weeks and were instructed on how to administer the trial product. During this period the subjects demonstrated that they could adhere to the injection regimen in the trial.
Groups:
- Liraglutide: Subjects received liraglutide once daily by subcutaneous injection in the abdomen, thigh or upper arm, at any time of the day and irrespective of meals, for a treatment period of 42 to 60 months. It was recommended to keep the time of injection consistent from day to day. Liraglutide was initiated at a dose of 0.6 mg and up-titrated to 1.2 mg after 1 week and to 1.8 mg after one additional week up to 42-60 months.
- Placebo: Subjects received placebo (matched to liraglutide) daily by subcutaneous injection in the abdomen, thigh or upper arm, at any time of the day and irrespective of meals, for a treatment period of 42 to 60 months. It was recommended to keep the time of injection consistent from day to day. Placebo was initiated at a dose of 0.6 mg and up-titrated to 1.2 mg after 1 week and to 1.8 mg after one additional week up to 42-60 months.
Period: Overall Study
Arm/Group | Liraglutide | Placebo
Started | 4668 | 4672
Completed | 4529 | 4513
Not Completed | 139 | 159
Not completed — Withdrawn - does not allow contact | 4 | 8
Not completed — Lost to Follow-up | 8 | 9
Not completed — Alive | 127 | 142

BASELINE CHARACTERISTICS:
Population: All the randomised subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Placebo | Total
Number analyzed (Participants) | 4668 | 4672 | 9340
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (7.2) | 64.4 (7.2) | 64.3 (7.2)
Age, Customized [Number; unit: Participants]
  Between 18 and 64 years | 2512 | 2499 | 5011
  Between 65 to 84 years | 2139 | 2148 | 4287
  85 years and over | 17 | 25 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1657 | 1680 | 3337
  Male | 3011 | 2992 | 6003

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomisation to First Occurrence of Cardiovascular Death, Non-fatal Myocardial Infarction, or Non-fatal Stroke (a Composite Cardiovascular Outcome)
Description: Time from randomisation to first occurrence of cardiovascular death, non-fatal myocardial infarction, or non-fatal stroke (a composite cardiovascular outcome). The percentage of subjects experiencing a first event of cardiovascular death, non-fatal myocardial infarction, or non-fatal stroke (a composite cardiovascular outcome) is presented.
Time Frame: from randomisation (visit 3; month 0) to last contact (visit 16; up to month 60+30 days)
Population: All randomised subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 4668 | 4672
percentage of subjects | 13.0 | 14.9
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; The primary endpoint was evaluated using the Cox regression model to estimate the hazard ratio (HR) (liraglutide/placebo) and the 2-sided 95% confidence interval (CI) including treatment group as factor. Non-inferiority of liraglutide versus placebo was considered confirmed, if the upper limit of the two-sided 95% CI for the hazard ratio was below 1.3 or if the p-value for the one-sided test of H0: HR >=1.3 against Ha: HR <1.3 was less than 2.5% (or equivalent to 5% in two-sided test); Test type: Non-Inferiority or Equivalence — Non-inferiority of liraglutide versus placebo was considered confirmed, if the upper limit of the two-sided 95% CI for the hazard ratio was below 1.3 or if the p-value for the one-sided test of H0: HR >=1.3 against Ha: HR <1.3 was less than 2.5% (or equivalent to 5% in two-sided test). If non-inferiority was established for the primary outcome, a test for superiority was to be performed; p < 0.001, Regression, Cox — p-value is reported for one-sided (α-level 0.025) test for non-inferiority (hazard ratio >=1.3); Hazard Ratio (HR) = 0.868, 95% CI 2-sided [0.778 to 0.968]
Statistical Analysis 2: Comparison: Liraglutide vs Placebo; If non-inferiority was established for the primary outcome, a test for superiority was performed. Superiority of liraglutide versus placebo was considered confirmed, if the upper limit of the two-sided 95% CI for the hazard ratio was below 1.0 or equivalent if the p-value for the one-sided test of H0: HR >=1.0 against Ha: HR <1.0 was less than 2.5% (or equivalent to 5% in two-sided test); Test type: Superiority or Other; p = 0.005, Regression, Cox — p-value is reported for one-sided (α-level 0.025) test for superiority (hazard ratio>=1.0); Hazard Ratio (HR) = 0.868, 95% CI 2-sided [0.778 to 0.968]

2. Secondary Outcome: Time From Rand. to First Occurrence of an Expanded Composite Cardiovascular Outcome Defined as Either Cardiovascular Death, Non-fatal Myocardial Infarction, Non-fatal Stroke, Revascularisation, Hospitalisation for Unstable Angina or for Heart Failure.
Description: Time from randomisation to first occurrence of an expanded composite cardiovascular outcome defined as either cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, coronary revascularisation, hospitalisation for unstable angina or for heart failure. The percentage of subjects experiencing first occurrence of an expanded composite cardiovascular outcome defined as either cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, coronary revascularisation, hospitalisation for unstable angina or for heart failure is presented.
Time Frame: from randomisation (visit 3; month 0) to last contact (visit 16; up to month 60+30 days)
Population: All randomised subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 4668 | 4672
percentage of subjects | 20.3 | 22.7
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; Regression, Cox; The analysis was done using a Cox regression model with treatment as a fixed factor including all randomised subjects; Hazard Ratio (HR) = 0.881, 95% CI 2-sided [0.807 to 0.962]

3. Secondary Outcome: Time From Randomisation to All Cause Death
Description: Time from randomisation to all cause death. The percentage of subjects with a death by any cause (all-cause death) is presented.
Time Frame: from randomisation (visit 3; month 0) to last contact (visit 16; up to month 60+30 days)
Population: All randomised subjects
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 4668 | 4672
percentage of subjects | 8.2 | 9.6
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; Regression, Cox; The analysis was done using a Cox regression model with treatment as a fixed factor including all randomised subjects; Hazard Ratio (HR) = 0.847, 95% CI 2-sided [0.739 to 0.971]

4. Secondary Outcome: Time From Randomisation to Each Individual Component of the Expanded Composite Cardiovascular Outcome
Description: Time from randomisation to each individual component of the expanded composite cardiovascular outcome. The percentage of subjects experiencing each of the individual component of the expanded composite cardiovascular outcome (defined as either cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, coronary revascularisation, hospitalisation for unstable angina or heart failure) is presented.
Time Frame: from randomisation (visit 3; month 0) to last contact (visit 16; up to month 60+30 days)
Population: All the randomised subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 4668 | 4672
percentage of subjects
  Cardiovascular death | 4.7 | 6.0
  Non-fatal stroke | 3.4 | 3.8
  Non-fatal myocardial infarction | 6.0 | 6.8
  Unstable angina pectoris (hospitalisation) | 2.6 | 2.7
  Coronary revascularisation | 8.7 | 9.4
  Heart failure (hospitalisation) | 4.7 | 5.3
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing cardiovascular death was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.783, 95% CI 2-sided [0.656 to 0.934]
Statistical Analysis 2: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing non-fatal stroke was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.894, 95% CI 2-sided [0.721 to 1.107]
Statistical Analysis 3: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing non-fatal myocardial infarction was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.878, 95% CI 2-sided [0.747 to 1.031]
Statistical Analysis 4: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing hospitalisation for unstable angina pectoris was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.980, 95% CI 2-sided [0.763 to 1.258]
Statistical Analysis 5: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing coronary revascularisation was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.912, 95% CI 2-sided [0.797 to 1.044]
Statistical Analysis 6: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing hospitalisation for heart failure was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.872, 95% CI 2-sided [0.727 to 1.046]

5. Secondary Outcome: Time From Randomisation to First Occurrence of a Composite Microvascular Outcome
Description: Time from randomisation to first occurrence of a composite microvascular outcome, defined as any one of the following:
  * new onset of persistent macroalbuminuria
  * persistent doubling of serum creatinine
  * need for continuous renal replacement therapy
  * death due to renal disease
  * need for retinal photocoagulation or treatment with intravitreal agents
  * vitreous haemorrhage
  * diabetes-related blindness
  The percentage of subjects experiencing a first occurrence of a composite microvascular outcome is presented.
Time Frame: from randomisation (visit 3; month 0) to last contact (visit 16; up to month 60+30 days)
Population: All randomised subjects.
Measure: Number; unit: Percentage of subjects
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 4668 | 4672
Percentage of subjects | 7.6 | 8.9
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing a first microvascular event was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.841, 95% CI 2-sided [0.730 to 0.969]

6. Secondary Outcome: Time From Randomisation to Each Individual Component of the Composite Microvascular Outcome and to the Retinopathy and Nephropathy Composite Outcomes Separately.
Description: Time from randomisation to each individual component of the composite microvascular outcome and to the retinopathy and nephropathy composite outcomes separately. The percentage of subjects experiencing each individual component of the composite microvascular outcome are presented.
Time Frame: from randomisation (visit 3; month 0) to last contact (visit 16; up to month 60+30 days)
Population: All randomised subjects
Measure: Number; unit: Percentage of subjects
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 4668 | 4672
Percentage of subjects
  Nephropathy composite | 5.7 | 7.2
  New onset of persistent macroalbuminuria | 3.4 | 4.6
  Persistent doubling of serum creatinine | 1.9 | 2.1
  Need for continuous renal-replacement therapy | 1.2 | 1.4
  Death due to renal disease | 0.2 | 0.1
  Retinopathy composite | 2.3 | 2.0
  Treatment with photocoagulation/intravitreal agent | 2.1 | 1.8
  Development of diabetes-related blindness | 0.0 | 0.02
  Vitreous haemorrhage | 0.7 | 0.5
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing a composite nephropathy event was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.782, 95% CI 2-sided [0.666 to 0.918]
Statistical Analysis 2: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing a new onset of persistant macroalbuminaria event was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.738, 95% CI 2-sided [0.602 to 0.905]
Statistical Analysis 3: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing persistent doubling of serum creatinine was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.890, 95% CI 2-sided [0.667 to 1.189]
Statistical Analysis 4: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing a need for continuous renal-replacement therapy was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.869, 95% CI 2-sided [0.607 to 1.244]
Statistical Analysis 5: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing death due to renal disease was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.593, 95% CI 2-sided [0.521 to 4.869]
Statistical Analysis 6: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing composite retinopathy was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.149, 95% CI 2-sided [0.869 to 1.519]
Statistical Analysis 7: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing treatment with photocoagulation or intravitreal agents was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.159, 95% CI 2-sided [0.869 to 1.546]
Statistical Analysis 8: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing development of diabetes-related blindness was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.335, 95% CI 2-sided [0.004 to 30.847]
Statistical Analysis 9: Comparison: Liraglutide vs Placebo; Analysis for percentage of subjects experiencing vitreous haemorrhage was done by Cox regression model with treatment as fixed factor; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.454, 95% CI 2-sided [0.845 to 2.502]

ADVERSE EVENTS:
Time Frame: Adverse events from randomisation (visit 3; month 0) and until follow up (visit 16; up to month 60+30 days of post-treatment follow-up).
Description: Safety was assessed using the full analysis set which included all randomised subjects.
  Serious adverse events were systematically collected. Non-serious adverse events included both systematically collected as well as non-systematically collected adverse events.
Arm/Group | Liraglutide | Placebo
Serious Adverse Events (participants affected / at risk) | 2320/4668 | 2354/4672
Other Adverse Events (participants affected / at risk) | 684/4668 | 210/4672
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=4668) | Placebo (N=4672)
Abdominal abscess (Infections and infestations) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 5 (5)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 20 (20) | 15 (16)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 4 (4)
Abdominal panniculectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (2) | 4 (5)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 5 (5) | 6 (6)
Abscess neck (Infections and infestations) | 1 (2) | 2 (2)
Abscess of salivary gland (Infections and infestations) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 4 (4)
Accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acid peptic disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acquired oesophageal web (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acquired phimosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Actinic elastosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 37 (41) | 54 (59)
Acute hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 108 (124) | 94 (105)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 7 (7)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 155 (176) | 187 (211)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 10 (13)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 22 (23) | 18 (21)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Adams-Stokes syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (15) | 11 (11)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Adhesion (General disorders) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Adverse drug reaction (General disorders) | 1 (1) | 1 (1)
Afferent loop syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Air embolism (Vascular disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (2) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1) | 1 (1)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Amaurosis (Eye disorders) | 2 (2) | 0 (0)
Ammonia increased (Investigations) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 5 (5) | 2 (2)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 31 (32) | 21 (22)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anal skin tags (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 1 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 93 (105) | 93 (106)
Angina unstable (Cardiac disorders) | 144 (179) | 151 (180)
Angioedema (Skin and subcutaneous tissue disorders) | 6 (8) | 7 (7)
Angiogram peripheral (Investigations) | 1 (1) | 0 (0)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Angioplasty (Surgical and medical procedures) | 7 (8) | 11 (12)
Angle closure glaucoma (Eye disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (6)
Ankle operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2)
Aortic aneurysm (Vascular disorders) | 8 (8) | 5 (5)
Aortic aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Aortic bypass (Surgical and medical procedures) | 2 (2) | 1 (2)
Aortic dissection (Vascular disorders) | 3 (3) | 0 (0)
Aortic occlusion (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 11 (11) | 7 (7)
Aortic surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic valve calcification (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 2 (2)
Aortic valve sclerosis (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 6 (6) | 10 (10)
Aphakia (Eye disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 8 (8) | 11 (11)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 10 (11) | 5 (5)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Arterial repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Arterial restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Arterial therapeutic procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriogram coronary (Investigations) | 0 (0) | 7 (7)
Arteriosclerosis (Vascular disorders) | 3 (3) | 5 (5)
Arteriosclerosis coronary artery (Cardiac disorders) | 7 (7) | 12 (12)
Arteriosclerotic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 2 (3)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (4)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 13 (14)
Arthritis (Musculoskeletal and connective tissue disorders) | 16 (17) | 5 (5)
Arthritis bacterial (Infections and infestations) | 2 (2) | 3 (4)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asbestosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 9 (10) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 14 (23)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atherectomy (Surgical and medical procedures) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 89 (113) | 97 (112)
Atrial flutter (Cardiac disorders) | 17 (20) | 16 (18)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 4 (4)
Atrioventricular block (Cardiac disorders) | 1 (1) | 4 (4)
Atrioventricular block complete (Cardiac disorders) | 10 (10) | 9 (9)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 5 (5) | 4 (4)
Atrioventricular dissociation (Cardiac disorders) | 1 (1) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Aural polyp (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Autoimmune uveitis (Eye disorders) | 1 (1) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 3 (3) | 2 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
B-cell unclassifiable lymphoma low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Back disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (14) | 20 (21)
Bacteraemia (Infections and infestations) | 5 (5) | 6 (6)
Bacterial food poisoning (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 2 (2)
Barrett's oesophagus (Gastrointestinal disorders) | 2 (2) | 5 (5)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (17) | 7 (7)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Basal ganglia stroke (Nervous system disorders) | 1 (1) | 0 (0)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 25 (25) | 23 (23)
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (5)
Bile duct stone (Hepatobiliary disorders) | 3 (3) | 1 (2)
Biliary adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Biliary cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 5 (5) | 2 (3)
Biliary fistula (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 3 (5) | 2 (3)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder diverticulum (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder dysplasia (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder hypertrophy (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 2 (2) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 3 (3) | 1 (1)
Bladder squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 2 (2) | 0 (0)
Blood alcohol increased (Investigations) | 0 (0) | 1 (1)
Blood calcitonin increased (Investigations) | 0 (0) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 6 (6) | 3 (3)
Blood glucose fluctuation (Investigations) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 8 (8) | 8 (11)
Blood iron decreased (Investigations) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 2 (2) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 3 (3)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 11 (11) | 11 (11)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 2 (2)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1) | 1 (1)
Breast abscess (Infections and infestations) | 0 (0) | 2 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 6 (6)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 15 (15) | 24 (25)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 11 (13) | 19 (21)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 1 (1)
Bundle branch block left (Cardiac disorders) | 2 (2) | 2 (2)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Buried penis syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 10 (10) | 9 (9)
Calculus urinary (Renal and urinary disorders) | 2 (2) | 2 (2)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 2 (2) | 0 (0)
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 20 (20) | 31 (31)
Cardiac death (General disorders) | 4 (4) | 6 (6)
Cardiac discomfort (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 115 (138) | 137 (201)
Cardiac failure acute (Cardiac disorders) | 9 (11) | 11 (12)
Cardiac failure chronic (Cardiac disorders) | 28 (28) | 25 (29)
Cardiac failure congestive (Cardiac disorders) | 121 (180) | 129 (176)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 3 (3)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 (1) | 1 (1)
Cardiac stress test abnormal (Investigations) | 0 (0) | 1 (1)
Cardiac valve abscess (Infections and infestations) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac valve rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 2 (2) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 15 (15) | 13 (15)
Cardiogenic shock (Cardiac disorders) | 4 (4) | 11 (11)
Cardiomegaly (Cardiac disorders) | 0 (0) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 3 (4)
Cardiopulmonary bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 3 (3) | 6 (6)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Cardiospasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 2 (2)
Cardiovascular evaluation (Investigations) | 2 (2) | 2 (2)
Cardiovascular event prophylaxis (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 2 (2) | 0 (0)
Carotid angioplasty (Surgical and medical procedures) | 5 (5) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 2 (2) | 0 (0)
Carotid artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 3 (3) | 2 (2)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 28 (30) | 16 (18)
Carotid artery stent insertion (Surgical and medical procedures) | 6 (6) | 2 (2)
Carotid endarterectomy (Surgical and medical procedures) | 19 (23) | 14 (14)
Carotid revascularisation (Surgical and medical procedures) | 6 (6) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 6 (7) | 4 (4)
Cataract (Eye disorders) | 24 (29) | 32 (35)
Cataract operation (Surgical and medical procedures) | 2 (4) | 0 (0)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cataract traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Catheterisation cardiac (Investigations) | 2 (2) | 2 (2)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cell death (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 37 (50) | 54 (61)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 0 (0)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebellar haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 2 (2)
Cerebellar ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 4 (4) | 5 (5)
Cerebral hypoperfusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 14 (14) | 20 (21)
Cerebral ischaemia (Nervous system disorders) | 3 (3) | 3 (3)
Cerebral revascularisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 3 (3) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 52 (56) | 65 (68)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 2 (2)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 3 (3) | 6 (6)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Chest pain (General disorders) | 53 (56) | 49 (52)
Chills (General disorders) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Cholangitis (Hepatobiliary disorders) | 2 (3) | 4 (4)
Cholangitis acute (Hepatobiliary disorders) | 4 (4) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 11 (11) | 12 (12)
Cholecystitis acute (Hepatobiliary disorders) | 35 (35) | 18 (19)
Cholecystitis chronic (Hepatobiliary disorders) | 8 (8) | 5 (5)
Cholecystitis infective (Infections and infestations) | 3 (3) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 44 (45) | 30 (30)
Cholera (Infections and infestations) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholesterol granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chondrosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chondrosarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chordae tendinae rupture (Cardiac disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
Chronic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 52 (60) | 52 (55)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Chronic lymphocytic leukaemia stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 50 (68) | 59 (82)
Chronic pigmented purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 4 (5) | 6 (6)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Citrobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 6 (6) | 3 (3)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Coarctation of the aorta (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 4 (4) | 3 (4)
Colitis (Gastrointestinal disorders) | 9 (9) | 4 (4)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (14) | 16 (18)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonoscopy (Investigations) | 0 (0) | 1 (1)
Colonoscopy normal (Investigations) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colostomy closure (Surgical and medical procedures) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 2 (3)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Completed suicide (Psychiatric disorders) | 1 (1) | 4 (4)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Confusional state (Psychiatric disorders) | 0 (0) | 9 (9)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 11 (11) | 7 (7)
Contrast media allergy (Immune system disorders) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Cor pulmonale (Cardiac disorders) | 0 (0) | 1 (2)
Cor pulmonale acute (Cardiac disorders) | 0 (0) | 1 (1)
Cor pulmonale chronic (Cardiac disorders) | 1 (1) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 1 (1)
Coronary angioplasty (Surgical and medical procedures) | 46 (56) | 39 (42)
Coronary arterial stent insertion (Surgical and medical procedures) | 110 (117) | 112 (136)
Coronary artery bypass (Surgical and medical procedures) | 84 (86) | 102 (105)
Coronary artery disease (Cardiac disorders) | 73 (77) | 87 (89)
Coronary artery insufficiency (Cardiac disorders) | 2 (2) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 16 (16) | 10 (10)
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 5 (5) | 10 (10)
Coronary artery stenosis (Cardiac disorders) | 20 (20) | 35 (36)
Coronary ostial stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 120 (144) | 132 (157)
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Culture urine positive (Investigations) | 1 (1) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 7 (7) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Dacryocystitis (Infections and infestations) | 0 (0) | 1 (1)
Deafness bilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Death (General disorders) | 55 (55) | 47 (47)
Decreased activity (General disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Deep brain stimulation (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 20 (23) | 10 (11)
Dehydration (Metabolism and nutrition disorders) | 30 (30) | 22 (22)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 3 (3)
Dementia (Nervous system disorders) | 3 (3) | 3 (3)
Dementia Alzheimer's type (Nervous system disorders) | 2 (2) | 0 (0)
Dementia with Lewy bodies (Nervous system disorders) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Dependence on respirator (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 9 (11) | 7 (7)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermoid cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Device battery issue (General disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 2 (3) | 4 (5)
Device leakage (General disorders) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 2 (2) | 5 (5)
Device occlusion (General disorders) | 2 (3) | 3 (3)
Device related infection (Infections and infestations) | 5 (5) | 3 (5)
Device related sepsis (Infections and infestations) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 11 (12)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 25 (28) | 43 (47)
Diabetic blindness (Eye disorders) | 1 (1) | 1 (1)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 66 (88) | 80 (94)
Diabetic foot infection (Infections and infestations) | 11 (12) | 9 (11)
Diabetic gangrene (Infections and infestations) | 1 (1) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 11 (12) | 7 (8)
Diabetic mononeuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 6 (7) | 11 (11)
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 9 (10) | 7 (12)
Diabetic retinal oedema (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 9 (9) | 15 (15)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (4) | 2 (2)
Diabetic vascular disorder (Vascular disorders) | 2 (2) | 1 (1)
Dialysis related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 11 (11)
Diarrhoea infectious (Infections and infestations) | 2 (2) | 0 (0)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dilatation atrial (Cardiac disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (2) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 2 (2) | 4 (4)
Diverticulitis (Infections and infestations) | 7 (8) | 13 (13)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 2 (2) | 7 (7)
Diverticulum intestinal (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 (2) | 1 (2)
Dizziness (Nervous system disorders) | 12 (12) | 6 (6)
Drowning (General disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 4 (4) | 1 (1)
Drug interaction (General disorders) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 2 (2) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 8 (8) | 6 (6)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 5 (5)
Duodenal ulcer perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 4 (4) | 2 (2)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 32 (36)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7)
Dysuria (Renal and urinary disorders) | 1 (1) | 3 (3)
ECG signs of myocardial ischaemia (Investigations) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 2 (2)
Electric shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 3 (3)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 5 (6) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Endarterectomy (Surgical and medical procedures) | 0 (0) | 3 (3)
Endocarditis (Infections and infestations) | 3 (3) | 4 (4)
Endocarditis enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 2 (2)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Endometrial hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Enterobacter pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1) | 1 (1)
Epididymitis ureaplasmal (Infections and infestations) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 4 (5) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Erysipelas (Infections and infestations) | 10 (11) | 14 (16)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Extradural abscess (Infections and infestations) | 2 (2) | 1 (1)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 4 (4) | 1 (1)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecalith (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 84 (94) | 81 (83)
Fat embolism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 6 (7) | 5 (5)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Femur fracture (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Fibrillary glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 8 (8) | 4 (6)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Follicle centre lymphoma, follicular grade I, II, III stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Follicle centre lymphoma, follicular grade I, II, III stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Frostbite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 2 (2)
Gallbladder abscess (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 1 (2)
Gallbladder empyema (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder perforation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 2 (2) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 10 (13) | 12 (14)
Gas gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric banding (Surgical and medical procedures) | 1 (1) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 4 (4) | 6 (6)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 5 (5) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 15 (16) | 13 (14)
Gastritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 4 (4) | 10 (10)
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 33 (34) | 31 (31)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 9 (9) | 4 (4)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 2 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 14 (17) | 21 (27)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (3) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 (11) | 12 (12)
Gastroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 3 (3)
Generalised oedema (General disorders) | 2 (2) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 2 (2) | 1 (1)
Genital prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Giant cell tumour of tendon sheath (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 3 (3)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 1 (2) | 0 (0)
Glomerulosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomus tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 1 (1)
Goitre (Endocrine disorders) | 8 (8) | 5 (5)
Gout (Metabolism and nutrition disorders) | 4 (8) | 6 (6)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Granuloma (General disorders) | 1 (1) | 1 (1)
Granulomatosis with polyangiitis (Vascular disorders) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Haemangioma of spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 5 (5)
Haematoma (Vascular disorders) | 1 (1) | 2 (2)
Haematoma infection (Infections and infestations) | 1 (2) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 7 (7) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 6 (6) | 3 (4)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (2) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 4 (5)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 10 (10) | 13 (13)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 4 (4)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hamartoma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 7 (7)
Heart rate decreased (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 3 (3) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (3) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 4 (4) | 6 (6)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 3 (3) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatopulmonary syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 2 (2) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 6 (6)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 5 (6) | 4 (4)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Human bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Human ehrlichiosis (Infections and infestations) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 5 (6) | 2 (2)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercorticoidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 34 (35) | 49 (52)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (10) | 15 (15)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 32 (36) | 25 (27)
Hypertensive cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 14 (18) | 12 (13)
Hypertensive emergency (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Hypertensive heart disease (Cardiac disorders) | 2 (2) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaldosteronism (Endocrine disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 44 (60) | 75 (92)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 2 (2)
Hypoglycaemic seizure (Nervous system disorders) | 2 (2) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 21 (24) | 28 (28)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (8) | 7 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 18 (18) | 16 (17)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 6 (6) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2 (2) | 4 (5)
IIIrd nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ileal gangrene (Infections and infestations) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 4 (4) | 7 (7)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 2 (2)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1)
Imaging procedure (Investigations) | 1 (1) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 5 (6) | 1 (1)
Impaired healing (General disorders) | 4 (4) | 2 (2)
Implantable defibrillator insertion (Surgical and medical procedures) | 2 (2) | 5 (5)
Implantable defibrillator replacement (Surgical and medical procedures) | 1 (1) | 1 (1)
Incarcerated hernia (General disorders) | 2 (2) | 1 (1)
Incarcerated hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incision site infection (Infections and infestations) | 1 (1) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Incorrect dose administered (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Infected bites (Infections and infestations) | 1 (1) | 2 (2)
Infected dermal cyst (Infections and infestations) | 1 (1) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 4 (5)
Infection (Infections and infestations) | 2 (2) | 7 (7)
Infectious colitis (Infections and infestations) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (4) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Inflammation of wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inflammatory marker increased (Investigations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 8 (8)
Inguinal hernia (Gastrointestinal disorders) | 12 (15) | 14 (14)
Inguinal hernia repair (Surgical and medical procedures) | 2 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Intermittent claudication (Vascular disorders) | 5 (7) | 3 (3)
Internal carotid artery kinking (Nervous system disorders) | 1 (2) | 0 (0)
Internal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
International normalised ratio decreased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 3 (3) | 6 (6)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 13 (14) | 23 (27)
Intervertebral discitis (Infections and infestations) | 2 (2) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 7 (9)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial lipoma (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 9 (9)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 9 (9) | 13 (13)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 2 (3)
Ischaemic cardiomyopathy (Cardiac disorders) | 3 (3) | 9 (9)
Ischaemic cerebral infarction (Nervous system disorders) | 2 (3) | 4 (4)
Ischaemic heart disease prophylaxis (Surgical and medical procedures) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 50 (54) | 54 (59)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 2 (2)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 4 (5) | 2 (6)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Keloid scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 2 (2) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Labile hypertension (Vascular disorders) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Lacunar infarction (Nervous system disorders) | 6 (7) | 8 (8)
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large granular lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 16 (16) | 13 (18)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Laryngeal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 5 (5) | 10 (10)
Left ventricular end-diastolic pressure increased (Investigations) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 3 (3) | 7 (7)
Left ventricular hypertrophy (Cardiac disorders) | 3 (3) | 3 (3)
Legionella infection (Infections and infestations) | 0 (0) | 1 (1)
Leriche syndrome (Vascular disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 11 (11) | 3 (3)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lipoma excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Liposarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 2 (2) | 2 (2)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Lividity (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Lobar pneumonia (Infections and infestations) | 15 (16) | 15 (15)
Local swelling (General disorders) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 7 (9) | 8 (8)
Loss of consciousness (Nervous system disorders) | 5 (6) | 7 (7)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 15 (16) | 15 (15)
Lumbar radiculopathy (Nervous system disorders) | 4 (4) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 11 (12) | 9 (9)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 5 (5)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 9 (10)
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (2) | 1 (1)
Macular fibrosis (Eye disorders) | 2 (2) | 4 (4)
Macular oedema (Eye disorders) | 1 (1) | 1 (1)
Macular rupture (Eye disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 4 (5)
Malaise (General disorders) | 0 (0) | 3 (3)
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 3 (3)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 6 (6)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 2 (2) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Mass (General disorders) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Medical device battery replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical device change (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 2 (2) | 0 (0)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Melanocytic hyperplasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 2 (2)
Meningitis pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Mental disorder (Psychiatric disorders) | 1 (2) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3) | 3 (4)
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Mesenteric artery embolism (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Metabolic disorder (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 6 (6) | 0 (0)
Metabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Metaplasia (General disorders) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 4 (4)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Microalbuminuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Microangiopathy (Vascular disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 4 (4)
Mitral valve calcification (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 3 (3) | 10 (10)
Mitral valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Mononeuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Mucinous breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 7 (7) | 9 (9)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple system atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Myocardial fibrosis (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 68 (71) | 84 (89)
Myocardial ischaemia (Cardiac disorders) | 27 (27) | 33 (35)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasopharyngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (9) | 9 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Necrobiosis lipoidica diabeticorum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Necrosis (General disorders) | 0 (0) | 1 (1)
Necrosis ischaemic (Vascular disorders) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 4 (4) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 26 (27) | 21 (22)
Nephropathy (Renal and urinary disorders) | 6 (6) | 13 (15)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 2 (2) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 2 (2)
Nervous system disorder (Nervous system disorders) | 0 (0) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neuritis cranial (Nervous system disorders) | 0 (0) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neurogenic shock (Vascular disorders) | 0 (0) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (2) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 45 (52) | 63 (73)
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 8 (8) | 11 (11)
Obesity surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 2 (2) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 6 (6) | 9 (10)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Oesophageal squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Open angle glaucoma (Eye disorders) | 1 (1) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 3 (3)
Optic nerve infarction (Eye disorders) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Orchitis (Infections and infestations) | 2 (2) | 2 (2)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 10 (10) | 8 (8)
Orthostatic intolerance (Nervous system disorders) | 1 (1) | 0 (0)
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 75 (80) | 64 (69)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 21 (27) | 23 (30)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 2 (3)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 2 (2) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian epithelial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pain (General disorders) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3) | 4 (4)
Pancreas divisum (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Pancreas infection (Infections and infestations) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 7 (7)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 2 (2) | 2 (2)
Pancreatic disorder (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatic enzymes increased (Investigations) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (3) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 18 (20) | 10 (11)
Pancreatitis acute (Gastrointestinal disorders) | 14 (14) | 19 (22)
Pancreatitis chronic (Gastrointestinal disorders) | 2 (2) | 2 (2)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 3 (3)
Papilloedema (Eye disorders) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Parapsoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Parathyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Paratracheal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 2 (2)
Parkinsonism (Nervous system disorders) | 1 (1) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic floor repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Penetrating atherosclerotic ulcer (Vascular disorders) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 3 (3) | 4 (4)
Percutaneous coronary intervention (Surgical and medical procedures) | 59 (71) | 57 (66)
Periarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Pericardial cyst (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 3 (3)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 5 (5)
Pericarditis uraemic (Cardiac disorders) | 1 (1) | 1 (1)
Perichondritis (Infections and infestations) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 24 (27) | 34 (38)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 2 (2) | 1 (1)
Peripheral artery angioplasty (Surgical and medical procedures) | 20 (25) | 27 (29)
Peripheral artery bypass (Surgical and medical procedures) | 11 (12) | 14 (19)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Peripheral artery stenosis (Vascular disorders) | 8 (9) | 12 (19)
Peripheral artery stent insertion (Surgical and medical procedures) | 7 (10) | 9 (10)
Peripheral artery thrombosis (Vascular disorders) | 4 (5) | 4 (5)
Peripheral circulatory failure (Vascular disorders) | 1 (1) | 0 (0)
Peripheral endarterectomy (Surgical and medical procedures) | 6 (7) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 13 (14) | 11 (12)
Peripheral nerve lesion (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral revascularisation (Surgical and medical procedures) | 29 (33) | 36 (47)
Peripheral swelling (General disorders) | 0 (0) | 3 (3)
Peripheral vascular disorder (Vascular disorders) | 10 (11) | 8 (9)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Peritoneal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 5 (6) | 6 (9)
Peritonitis bacterial (Infections and infestations) | 3 (3) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Personality disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Peyronie's disease (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Phlebosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasmodium falciparum infection (Infections and infestations) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 15 (18)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 133 (154) | 141 (157)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (7)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia influenzal (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia viral (Infections and infestations) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumopericardium (Cardiac disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Polyneuropathy (Nervous system disorders) | 2 (2) | 2 (2)
Polyp (General disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Post procedural hypothyroidism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 6 (6) | 3 (3)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic headache (Nervous system disorders) | 1 (2) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Postoperative wound infection (Infections and infestations) | 9 (9) | 6 (6)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 6 (7) | 6 (6)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Proctitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Prophylaxis against dehydration (Surgical and medical procedures) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 (24) | 39 (39)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Prostatic dysplasia (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 7 (7) | 2 (2)
Prostatomegaly (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2) | 3 (3)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 2 (2)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 24 (26)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (8)
Pulmonary mycosis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 17 (22) | 21 (25)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 3 (3)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 9 (9) | 10 (12)
Pyelonephritis acute (Infections and infestations) | 6 (9) | 6 (6)
Pyrexia (General disorders) | 5 (6) | 6 (6)
Pyuria (Infections and infestations) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Reactive gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 6 (7) | 5 (6)
Rectal polyp (Gastrointestinal disorders) | 3 (3) | 2 (2)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 1 (1)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rehabilitation therapy (Surgical and medical procedures) | 1 (1) | 1 (1)
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 2 (2) | 3 (3)
Renal artery stent placement (Surgical and medical procedures) | 0 (0) | 3 (3)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Renal cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal cyst (Renal and urinary disorders) | 5 (5) | 11 (11)
Renal failure (Renal and urinary disorders) | 20 (21) | 31 (33)
Renal function test (Investigations) | 1 (1) | 0 (0)
Renal haemorrhage (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 14 (14) | 10 (10)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal revascularisation surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 5 (5)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 19 (21)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 7 (10)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Retinal aneurysm (Eye disorders) | 1 (1) | 0 (0)
Retinal artery embolism (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 2 (2) | 1 (1)
Retinal degeneration (Eye disorders) | 1 (1) | 1 (1)
Retinal detachment (Eye disorders) | 2 (2) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Retinal infarction (Eye disorders) | 2 (2) | 0 (0)
Retinal vascular occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 3 (4) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 2 (2) | 4 (5)
Retinopathy haemorrhagic (Eye disorders) | 1 (1) | 0 (0)
Retinopathy proliferative (Eye disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Retroperitoneal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhythm idioventricular (Cardiac disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Right ventricular failure (Cardiac disorders) | 0 (0) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 20 (23) | 16 (16)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salmonella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 2 (2) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 4 (4) | 3 (3)
Scrotal abscess (Infections and infestations) | 3 (3) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Seizure (Nervous system disorders) | 7 (7) | 6 (6)
Seizure like phenomena (Nervous system disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 48 (50) | 34 (36)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 8 (9) | 13 (13)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Serotonin syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Serum ferritin decreased (Investigations) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 5 (5) | 0 (0)
Short-bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Shunt occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Silent myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Single functional kidney (Renal and urinary disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 6 (6)
Sinus node dysfunction (Cardiac disorders) | 10 (10) | 9 (9)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin graft (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 10 (10) | 15 (15)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (7)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 10 (12) | 5 (23)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Social stay hospitalisation (Social circumstances) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 3 (3) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Somatisation disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Spinal claudication (Nervous system disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 7 (7) | 10 (10)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Spinal cord injury thoracic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 8 (8)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Splenic embolism (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 2 (2)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 2 (2) | 5 (5)
Staphylococcal sepsis (Infections and infestations) | 4 (4) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Steal syndrome (Vascular disorders) | 0 (0) | 1 (1)
Stent placement (Surgical and medical procedures) | 3 (3) | 4 (4)
Stent-graft endoleak (General disorders) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 4 (4) | 3 (3)
Subclavian artery stenosis (Vascular disorders) | 2 (2) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 5 (6) | 10 (10)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Subgaleal haematoma (Vascular disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 4 (4) | 6 (6)
Sudden death (General disorders) | 11 (11) | 17 (17)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 4 (4) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 9 (9) | 7 (9)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 39 (43) | 26 (27)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 2 (2) | 2 (2)
Systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (4) | 3 (3)
Tendon rupture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Testicular abscess (Infections and infestations) | 1 (1) | 0 (0)
Testicular cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular necrosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 3 (3) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Thrombectomy (Surgical and medical procedures) | 0 (0) | 4 (5)
Thromboangiitis obliterans (Vascular disorders) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 3 (4) | 0 (0)
Thrombosis (Vascular disorders) | 1 (2) | 0 (0)
Thrombosis in device (General disorders) | 1 (2) | 1 (1)
Thrombotic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 3 (3) | 0 (0)
Thyroid C-cell hyperplasia (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis subacute (Endocrine disorders) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 5 (5)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 1 (1) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 2 (3)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 3 (4)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 52 (57) | 68 (73)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 3 (3)
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transplant evaluation (Investigations) | 0 (0) | 1 (1)
Traumatic arthritis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic arthrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 4 (4)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis of genitourinary system (Infections and infestations) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 3 (3)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ulnocarpal abutment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 6 (6) | 4 (4)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3)
Uraemic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Ureteral necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteral polyp (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 4 (4) | 6 (7)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 8 (8) | 12 (13)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 47 (51) | 71 (79)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 3 (3)
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Urine albumin/creatinine ratio increased (Investigations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 8 (8) | 17 (19)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 6 (6)
Uterine prolapse (Reproductive system and breast disorders) | 3 (3) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 3 (3) | 5 (6)
Vaginal abscess (Infections and infestations) | 1 (1) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (2) | 2 (2)
Vascular dementia (Nervous system disorders) | 1 (1) | 2 (2)
Vascular graft (Surgical and medical procedures) | 1 (1) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 3 (3) | 6 (7)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Vascular operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Vasculitis necrotising (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 3 (3) | 0 (0)
Ventricular dyssynchrony (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 5 (5) | 3 (3)
Ventricular fibrillation (Cardiac disorders) | 4 (4) | 6 (6)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 18 (29) | 8 (11)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 6 (6) | 10 (10)
Vertigo positional (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 3 (3)
Viral infection (Infections and infestations) | 5 (5) | 2 (2)
Viral myocarditis (Infections and infestations) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 3 (3)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitreous adhesions (Eye disorders) | 2 (2) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 6 (6) | 5 (5)
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 17 (20) | 11 (11)
Vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Walking disability (Social circumstances) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 3 (3)
Weight increased (Investigations) | 0 (0) | 1 (1)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (4) | 2 (2)
Wound decomposition (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 6 (6) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound sepsis (Infections and infestations) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Wrong drug administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Zygomycosis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=4668) | Placebo (N=4672)
Diarrhoea (Gastrointestinal disorders) | 266 (355) | 102 (124)
Nausea (Gastrointestinal disorders) | 517 (655) | 129 (149)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.